CLINICAL TRIAL: NCT02283632
Title: A Trial of the Jejunal Diversion Procedure (Side-to-side Jejuno-jejunostomy) (Europe)
Brief Title: A Trial of the Jejunal Diversion Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESC-14-001
Record Dates: First submitted 2014-10-31; First posted 2014-11-05 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Jejunal Diversion (Experimental): all subjects who receive jejunal diversion surgery
  Interventions: Procedure: Jejunal Diversion

INTERVENTIONS:
Procedure: Jejunal Diversion — The jejuno-jejunostomy surgical procedure is a well-known general surgical operation performed for multiple acute and chronic conditions including Crohn's disease, ovarian cancer, and small bowel obstruction. The jejunal diversion procedure is an adaptation of a jejuno-jejunostomy. The proximal end of the anastomosis is approximately 100 cm distal from the ligament of Treitz. The distal end of the anastomosis is approximately 250 cm proximal from the ileocecal junction.

SUMMARY:
This is a single site trial to assess metabolic effects in subjects after a Jejunal Diversion procedure was performed.

DETAILED DESCRIPTION:
The Jejunal Diversion procedure is an adaptation of a jejuno-jejunostomy, which is a surgical procedure often used to address a mix of pathological conditions. The safety of the Jejunal Diversion procedure is not in question, but rather understanding the gastrointestinal signalling effects. Up to 25 eligible subjects will be enrolled into the trial. Enrollment will stop once 15 subjects have undergone the Jejunal Diversion procedure

ELIGIBILITY:
Inclusion Criteria:

1. 20 to 60 years of age (inclusive) on the date the ICD is signed
2. A BMI ≥ 27 kg/m2 and < 40 kg/m2
3. HbA1c ≥ 8% (63.9 mmol/mol) and ≤ 11% (96.7 mmol/mol)
4. C-peptide ≥ 3 ng/mL (0.999 nmol/L)
5. At least one of the following:

   1. Systolic BP ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg, or on anti-hypertensive medication
   2. HDL < 40 mg/dL (1.0344 mmol/L) (men) or < 50 mg/dL (1.293 mmol/L) (women), or on medication for low HDL
   3. LDL > 100 mg/dL (2.586 mmol/L), or on medication for high LDL
   4. TG ≥ 150 mg/dL (1.694 mmol/L) or on TG lowering medication treatment
   5. FPG ≥ 100 mg/dL (5.556 mmol/L) or on medication for hyperglycemia or anti-T2DM
6. Able to comprehend and sign the EC-approved trial ICD

Exclusion Criteria:

1. Unable or unwilling to attend follow-up visits and examinations
2. History of drug and/or alcohol abuse within 2 years of Screening Visit
3. Any previous major GI surgery (e.g., any GI surgery with a resection, etc.) Examples of previous GI surgery allowed include: appendectomy, gall bladder surgery, liver biopsies, endoscopic procedures, etc.
4. Scheduled concurrent surgical procedure
5. Women of childbearing potential who are pregnant or lactating at the time of screening, at the time of surgery, or planning to become pregnant during the follow-up period
6. Psychiatric disorders that may affect compliance with the clinical trial, including dementia, active psychosis, severe depression, or history of suicide attempts
7. Any condition which precludes compliance with the trial, including:

   1. Inflammatory diseases of the GI tract, including severe intractable esophagitis, gastric ulceration, duodenal ulceration, or specific inflammation such as Crohn's disease or ulcerative colitis that have been active within the past 10 years
   2. History of Hepatitis B or C
   3. T1DM
   4. LADA (confirmed by positive GAD autoantibodies, IAA, and ICA)
   5. Immunocompromised such as that resulting from chronic oral steroid use, cancer chemotherapeutic agents, or immune deficiency disorders
8. Screening laboratory tests with any of the following:

   1. ALT and/or AST levels ≥ 4 times ULN according to laboratory normal ranges
   2. Blood creatinine level ≥ 1.5 times ULN according to laboratory normal ranges
   3. BUN level ≥ 1.5 times ULN according to laboratory normal ranges
9. Use of any of the following medications in the past 120 days:

   1. Chronic steroid use
   2. Prescription or over-the-counter medications or supplements with a primary indication known to cause or assist in weight reduction
10. Use of any of the following medications in the past 60 days:

    a. Promotility agents
11. Any other medical condition or finding for which, at the discretion of the PI, the subject should be excluded
12. Participation in any other clinical trial (not to include registries or survey-only studies) within 30 days or 5 half lives of an investigational drug (which ever is longer), of Visit 1 (Screening Visit) and for the duration of the trial

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Assess change in glycosylated hemoglobin A1c | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robin Scamuffa, Study Director — Ethicon, Inc.
Locations (1):
- OB KlINIKA, Prague, Czechia

REFERENCES:
- [Derived] Fried M, Dolezalova K, Chambers AP, Fegelman EJ, Scamuffa R, Schwiers ML, Waggoner JR, Haluzik M, Seeley RJ. A novel approach to glycemic control in type 2 diabetes mellitus, partial jejunal diversion: pre-clinical to clinical pathway. BMJ Open Diabetes Res Care. 2017 Sep 1;5(1):e000431. doi: 10.1136/bmjdrc-2017-000431. eCollection 2017. PMID 29225893